CLINICAL TRIAL: NCT04711642
Title: Comprehensive Study on Dry Eye and Ocular Surface Disease Prior and After Cataract Surgery: Effects of Treatment on Dry Eye and Inflammatory Biomarkers.
Brief Title: Comprehensive Study on Dry Eye and Ocular Surface Disease Prior and After Cataract Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Oftalmológica Los Andes (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dry Eye and Cataract Surgery
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye Disease; Dry Eye Syndrome; Evaporative Dry Eye; Cataract; Phacoemulsification
Keywords: Cataract surgery; Dry eye disease; Ocular surface osmolarity; matrix metalloproteinase-9
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Intervention Model Description: Eligible patients will be enrolled and randomly assigned by a computer generated randomization list in a 1:1:1 ratio to the intervention groups (2) or the control group. After cataract surgery, all groups will be given a topical steroid-antibiotic (tobramycin 0.3% and dexamethasone acetate 0.1%) commercially available and commonly used by ophthalmologists worldwide postoperatively, in a 3-week tapered regimen (every 2 hours the first day, then every 4 hours for 6 days, then 3 times a day for 1 week and twice a day for 1 week). The 2 study groups will be also prescribed lubricant eye drops from the postoperative day 7 containing sodium hyaluronate 0.1% (in 2 different commercially available formulations) to instill 4 times daily for the following 3 months. Study group patients will be instructed to instill the lubricant eyedrops at least 10 minutes after the tobramycin-dexamethasone eyedrops. At postoperative visits, patients will be asked about compliance with the assigned treatment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- No intervention (No Intervention): Control group.
- Treatment 1 (Experimental): Sodium hyaluronate 0.1% eyedrops (Systane ultra plus), q.i.d from day 7 to day 30 after cataract surgery.
  Interventions: Drug: The study will include three arms, one non interventional and 2 interventions. The intervention arms will include two commercially available sodium hyaluronate 0.1% (Systane ultra plus and Hylo-comod)
- Treatment 2 (Experimental): Sodium hyaluronate 0.1% eyedrops (Hylo-comod), q.i.d from day 7 to day 30 after cataract surgery.
  Interventions: Drug: The study will include three arms, one non interventional and 2 interventions. The intervention arms will include two commercially available sodium hyaluronate 0.1% (Systane ultra plus and Hylo-comod)

INTERVENTIONS:
Drug: The study will include three arms, one non interventional and 2 interventions. The intervention arms will include two commercially available sodium hyaluronate 0.1% (Systane ultra plus and Hylo-comod) — All groups will receive a topical steroid-antibiotic for 3 weeks. The study groups will be also prescribed eye drops containing sodium hyaluronate 0.1% from the postoperative day 7 for 4 weeks.
  Arms: Treatment 1; Treatment 2

SUMMARY:
Ocular surface disease (OSD), particularly dry eye, is one of the most common conditions seen by ophthalmologists. Dry eye (DE) is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear instability. DE significantly reduces quality of life and affects 5-30% of the population. As the proportion of individuals over age 60 increases because of greater life expectancies, we can anticipate the number of people with dry eye will also increase, which represents a major challenging for aging societies, like the Chilean one.

In the last few years clinical research on OSD is being intensely focused on diagnostic criteria, treatment strategies, methods used in diagnosis and better correlations between symptoms and clinical test results. All these lines of interest aim to improve the understanding of alterations and consequences occurring in the ocular surface disorders. Diagnostic testing is greatly valuable both for the detection of early changes due to DE and also to grade the severity of surface disease. The most commonly performed tests include the Schirmer test, tear break up time (TBUT), and ocular surface staining. However, newer point-of-care diagnostics tests such as tear osmolarity and matrix metalloprotease-9 (MMP-9) have been shown to have a high sensitivity and specificity in diagnosing ocular surface dysfunction.

Given that ocular surface dysfunction has been shown to have an adverse impact on visual function and can worsen after surgery, it is critical to identify and address any tear film and ocular surface abnormalities before cataract surgery. In the setting of preoperative cataract surgery planning, DE disease and meibomian gland dysfunction can impair critical refractive measures such as keratometry values worsening surgical outcomes.

To the best of our knowledge there are no ongoing or published studies that have evaluated DE and OSD as evidenced by either an abnormal tear-film parameter (elevated MMP-9 or abnormal osmolarity), or corneal surface and meibography evaluation findings (using novel non-invasive technology) in patients previous and after cataract surgery.

DETAILED DESCRIPTION:
A prospective randomized study has been designed to assess and characterize OSD/DE in consecutive patients presenting for cataract surgery evaluation and to identify eventual changes on biomarkers of the tear film of the same population postoperatively. At the same time, 2 different postoperative eye drops regimen will be evaluated in order to determine its impact on postoperative OSD/DE.

All group of patients will be subjected to Dry Eye assessment using diagnosis criteria and methodologies recommended by the 2017 Dry Eye Workshop (DEWS II) (2), which includes the assessment of a battery of symptoms (OSDI questionnaire), signs (tear meniscus height, corneal and conjunctival lissamine green/fluorescein staining), laboratory tests (Schirmer I, TBUT assessment, tear osmolarity, tear MMP-9, meibography, ocular redness, lipid layer thickness) and physical examination (lid, meibum gland assessment). This assessment will be carried out in all groups preoperative and at postoperative week 4 and postoperative week 12.

Altogether, by identifying definite changes either in novel tear film biomarkers or non invasive ocular tests of patients subjected to cataract surgery, we expect to contribute to the understanding of the pathophysiology of the OSD and Dry Eye associated to cataract surgery and to give lights on the utility of those changes as biomarkers in diagnosis and therapy assessment in these conditions committing the ocular surface.

The research hypothesis is that there is a high prevalence of ocular surface dysfunction among patients presenting for cataract surgery as measured by point-of-care objective tear tests and cataract surgery results in altered ocular surface in a major fraction of patients. Dry eye symptoms are not necessary associated with objective signs in the ocular surface, but are less in the group of patients treated with associated lubricant eyedrops postoperatively. Patients more symptomatic in the postoperative period tend to have multiple preoperative OSD/DE biomarkers altered.

Consecutive patients presenting for cataract surgery evaluation will be recruited at the Fundacion Oftalmologica Los Andes (FOLA) Ophthalmology Clinic (Santiago, Chile). Patients will be eligible according to inclusion and exclusion criteria indicated. Eligible patients will be invited to participate voluntary in the study. The study will comprise three groups with 30-35 patients per group. Dry eye patients will be diagnosed according to TFOS DEWS II report and to the recommendations of the Dry Eye Workshop of 2017. It will basically consist of: a) patient history: symptoms and signs (e.g. ocular irritation, dryness or foreign body sensation, redness, etc), exacerbating conditions, duration of symptoms, etc., will be obtained by using the Ocular Surface Disease Index (OSDI). b) physical examination: visual acuity measurement, external examination and slit lamp biomicroscopy (tear film, tear meniscus, eyelashes, eyelid margins, conjunctiva, cornea, lens and retina). c) Diagnostic tests: Tear film osmolarity (using Tearlab), Tear film MMP-9 levels (using InflammaDry). Non-invasive tests will be performed using Keratograph 5M, which includes: non-invasive tear film break up time tear meniscus height, lipid layer thickness, ocular redness and meibography.

The study will comprise three groups. Each group will comprise 30-35 patients. Each of the 100 patients will be featured by a list of clinical parameters (ocular signs and symptoms and laboratory tests used conventionally for Dry Eye diagnostic). It is expected to observe differences in parameters before and after cataract surgery and between the control group and the two interventional groups. Association of those differences with the type of postoperative regimen will be defined statistically by using Student t-test and ANOVA for parametric data and U-test of Mann-Whitney for non-parametric data (p<0.05 will be taken as significant). Altogether, it is expected that such a multiplicity of signs and symptoms will give valuable data on specificities of Dry Eye after cataract surgery.

All the participant surgeons will have a summary document of the inclusion and exclusion criteria and a flowchart of the patient's enrollment process to improve compliance. The data will be stored on an external digital platform and only the data analyst will have access to it. In addition, there will be written records of each enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Indication of phacoemulsification for refractive purposes or for the presence of visually significant cataract.
* Absence of intraoperative or postoperative complications of phacoemulsification
* Willing to participate in the study (signed informed consent)

Exclusion Criteria:

* Ocular surgeries within the previous 6 months.
* Contact lenses user.
* Severe blepharitis.
* Palpebral malposition and secondary dry eye
* History of filamentary keratitis, corneal neovascularization, or herpetic keratitis within previous 3 months.
* Hypersensitivity to investigated substances or diagnostic stains used.
* Antiglaucomatous topical medication
* Artificial tears with instillation frequency greater than 3 times a day in the last week

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Dry eye ocular symptoms | Baseline, 30 days, 90 days
  Difference in Ocular Surface Disease Index (OSDI) scores between groups.

SECONDARY OUTCOMES:
Non-invasive Break-up time | Baseline, 30 days, 90 days
  Difference in NIBUT scores between treated and untreated groups and between treated groups using 2 different lubricating drops.
Tear osmolarity | Baseline 30 days, 90 days
  Difference in Tear Osmolarity between treated and untreated groups and between treated groups using 2 different lubricating drops.
InflammaDry (MMP9) test | Baseline, 30 days, 90 days
  Difference in proportion of patients with a positive InflammaDry (MMP9) between treated and untreated groups and between treated groups using 2 different lubricating drops.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Montecinos Buneder, MD, Principal Investigator — Fundacion Oftalmologica Los Andes; Juan Stoppel Ortiz, MD, Principal Investigator — Fundacion Oftalmologica Los Andes; Felipe Valenzuela Santana, MD, Study Chair — Fundación Oftalmológica Los Andes; Cristobal Loezar Hernandez, MD, Principal Investigator — Fundacion Oftalmologica Los Andes

IPD SHARING:
Plan to Share IPD: No